CLINICAL TRIAL: NCT01974583
Title: Wound-healing Improvement by Resurfacing Split-Thickness Skin Donor Sites With Thin Split-thickness Grafting
Status: Completed | Type: Observational
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Principal Investigator, Yongqian Bian, Mr Yongqian Bian, Tang-Du Hospital
Other Study IDs: TDLL-2030130
Record Dates: First submitted 2013-09-12; First posted 2013-11-01 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Skin Graft Disorder; Disorder of Skin Donor Site; Wound Healing Disturbance of
Keywords: the split-thickness skin graft （STSG） donor site; regraft; wound healing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- the treatment group A: The people in treatment group were regrafted with thin split-thickness skin graft
  Interventions: Procedure: regrafted with thin split-thickness skin graft
- the control group B: The group B covered with the occlusive hydrocellular dressing (Allevyn Adhesive, Smith & Nephew)
  Interventions: Procedure: covered with the occlusive hydrocellular dressing
- the control group C: Group C were covered with paraffin gauze
  Interventions: Procedure: covered with paraffin gauze

INTERVENTIONS:
Procedure: regrafted with thin split-thickness skin graft — Group A (the treatment group) were regrafted with thin split-thickness skin graft
  Groups: the treatment group A
Procedure: covered with the occlusive hydrocellular dressing — group B covered with the occlusive hydrocellular dressing (Allevyn Adhesive, Smith & Nephew)
  Groups: the control group B
Procedure: covered with paraffin gauze — Group C covered with paraffin gauze
  Groups: the control group C

SUMMARY:
Split-thickness skin grafting remains fundamental treatment of patients with deep burns and other traumatic injuries. However, the split-thickness skin graft (STSG) donor site dressing has been controversial until now. Our study here aimed to assess patient comfort and wound-healing efficacy with the application of thin split-thickness grafting on STSG donor sites.

DETAILED DESCRIPTION:
Background：Split-thickness skin grafting remains fundamental treatment of patients with deep burns and other traumatic injuries. However, the split-thickness skin graft (STSG) donor site dressing has been controversial until now. Our study here aimed to assess patient comfort and wound-healing efficacy with the application of thin split-thickness grafting on STSG donor sites.

Methods: 192 consecutive patients undergoing split-thickness skin grafting were included in the study and the participants were randomly divided into three groups: Group A was regrafted with thin STSG, while, Group B and Group C were covered with the occlusive hydrocellular dressing and paraffin gauze, respectively. The three groups were compared regarding to the time of epithelialization, pain sensed by the patients and the scar formation.

ELIGIBILITY:
Inclusion Criteria:

* patients who continuously received an STSG from January 2002 to December 2010 in Department of Burn and Plastic Surgery, Tangdu Hospital, Fourth Military Medical University

Exclusion Criteria:

* The patients who were significant psychiatric, hypersensitive to silver, and not be followed up were excluded

Ages: 5 Years to 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study cohort included 192 participants, who were randomly selected from patients who continuously received an STSG from January 2002 to December 2010 in Department of Burn and Plastic Surgery, Tangdu Hospital, Fourth Military Medical University.
Sampling Method: Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2002-01; Primary Completion 2010-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
The time of epithelialization | up to 4 weeks
  The time of epithelialization was observed every 3 days

SECONDARY OUTCOMES:
Pain sensed by the patients | up to 6 months
  Pain sensed by the patients was assessed by Wong-Baker FACES Pain Rating Scale on day 2 and 5 after surgery

OTHER OUTCOMES:
Scar formation of skin donor site | 1 year
  Scar formation of skin donor sites was evaluated by Vancouver scar scale in terms of colour, vascular distribution, thickness and scratchability 6-12 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yongqian Bian, doctor, Study Director — specify Unaffiliated